CLINICAL TRIAL: NCT05103956
Title: Regular Treatment Versus Hemostatic Patch/Collagen Sealant and Polyethylene Glycol (Hemopatch) in the Immediate Postoperative of the Thyroidectomy, Unicentric Study, Non-inferiority, Open and Randomized (Tiropatch Study)
Brief Title: Hemostatic Patch/Collagen Sealant and Polyethylene Glycol (Hemopatch) in the Postoperative of the Thyroidectomy.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: TIROPATCH
Record Dates: First submitted 2021-10-07; First posted 2021-11-02 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-10

CONDITIONS: Goiter
MeSH Terms: conditions — Goiter

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A (Study Group): HEMOPATCH® (Sealing / hemostatic patch of collagen and e polyethylene glycol)
- Group B (Control Group): No hemostatic or the standard (ligatures and oxidized cellulose regenerated).

SUMMARY:
Observational study with non-inferiority, prospective, randomized (1: 1) and open-label medical device. The study has 2 treatment groups (HEMOPATCH® versus standard hemostasis).

DETAILED DESCRIPTION:
The main objective is to determine if there is a reduction in the volume of exudate in the surgical bed with the application of the collagen and polyethylene glycol hemostatic agent.

The present study includes patients undergoing total thyroidectomy for multinodular goiter in the Endocrine Surgery Unit of the Virgen del Rocío University Hospital.

The estimated sample calculation of patients enrolled in the study is 108 (2 groups, 1:1 ratio).

The patients don´t know what type of hemostatic the patients are going to receive (single blind).

The duration of patient follow-up will be 30 +/- 10 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients of legal age.
* Indication of total thyroidectomy due to multinodular goiter.
* Accept to enter the study and sign the informed consent.
* Patient willing and able to complete clinical trial procedures, as described described in the protocol.

Exclusion Criteria:

* Patients under 18 years of age.
* Patients with surgical indication for hemithyroidectomy or subtotal thyroidectomy (eg unilateral nodular goiters).
* Multinodular goiter with high suspicion or preoperative diagnosis of cancer (Bethesda V and VI and / or infiltration of neighboring structures on imaging tests).
* Known allergy or hypersensitivity to a component of the Hemopatch® investigational treatments, riboflavin, or bovine proteins.
* Concurrent or prior therapy with systemic pharmacological agents that promote blood clotting, including, but not limited to, tranexamic acid, activated factor VII, fibrinogen, and aprotinin.
* Pregnancy or breastfeeding.
* Refuse to enter the study and sign the informed consent.
* Not agreeing to carry out all the planned follow-up.
* Concurrent participation in another clinical trial with a medical device or drug or with interfering endpoints Inability to understand the nature and scope of the trial and the required procedures.

Criteria to be verified during surgery (Intraoperative exclusion criteria):

* Persistent major bleeding after primary hemostasis.
* Infection of the surgical area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The present study includes older patients who underwent total thyroidectomy for multinodular goiter in the Endocrine Surgery Unit of the Virgen del Rocío University Hospital. They must sign an informed consent and know the study procedures that are detailed in the protocol.
Sampling Method: Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Rate of changes in the exudate volume of the surgical bed with the application of the hemostatic agent of collagen and polyethylene glycol. | Up to 18 hours.
  Fixed periods of time will be established to evaluate the exudate from the surgical bed.
  It will be evaluated 18 hours after surgery by cervical ultrasound.

SECONDARY OUTCOMES:
Rate of changes in the patient's symptoms in the postoperative period of thyroidectomy after the application of the hemostatic agent of collagen and polyethylene glycol. | Up to 4 weeks.
  Decrease in the number of dyspnea at 24 hours and 30 days postoperatively.
Improvement in patient satisfaction after the application of the collagen and polyethylene glycol hemostatic agent, in relation to the surgical experience in the postoperative period of thyroidectomy. | Up to 4 weeks.
  Satisfaction survey at discharge and 30 days after the intervention.
Rate of improvement in postoperative complications of thyroidectomy after the application of the collagen and polyethylene glycol hemostatic agent. | Up to 4 weeks.
  Performance of the Trousseau test every 8 hours from surgery to hospital discharge and Calcemia (mg/dl) at discharge and at check-up in consultations (30 days) with total proteins.
Incidence rate of adverse effects after the use of the collagen and polyethylene glycol hemostatic agent in thyroid surgery. | Up to 24 weeks.
  Number of adverse events that have occurred in study patients.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Manuel Martos Martínez, Principal Investigator — Hospitales Universitarios Virgen del Rocío
Locations (1):
- Hospital Universitario Virgen del Rocío, Seville, Spain